CLINICAL TRIAL: NCT02000336
Title: Comparison of the Efficacy and Safety of Two Different Starting Dosages of Prednisolone in Early Active Rheumatoid Arthritis: a Randomized, Placebo Controlled Trial
Brief Title: Comparison of the Effectiveness of Two Different Dosages of Cortisone Compared to Placebo in Rheumatoid Arthritis
Acronym: CORRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prof. Dr. rer. nat. H.J. Trampisch (Other)
Collaborators: Ruhr University of Bochum (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. rer. nat. H.J. Trampisch, Professor Dr. rer.nat., Ruhr University of Bochum
Organization: Ruhr University of Bochum (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01KG1204; 2012-004074-25 (EudraCT Number)
Record Dates: First submitted 2013-11-19; First posted 2013-12-04 (Estimated); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Progression of Rheumatoid Arthritis
Keywords: radiographic damage; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Prednisolone; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Prednisolone 10 (Experimental): Prednihexal (Prednisolon), daily oral tablet, 10 mg during week one to four, 7,5 mg during week five to eight. Finally 5 mg for four weeks.
  Interventions: Drug: Prednisolone
- Prednisolone 60 (Experimental): Prednihexal (Prednisolon), daily oral tablet, 60 mg during the first week, weekly tapering: 40 mg, 20mg, 15mg, 10mg, 7,5mg. 7,5mg continued for one more week. Finally 5 mg for four weeks
  Interventions: Drug: Prednisolone
- Placebo (Placebo Comparator): daily oral tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisolone — To compare two standard p.o. GC starting dosages and the non-use of GCs in the treatment of patients with early active RA on the background of the established 'anchor' therapy with methotrexate (MTX).
  Other Names: PredniHexal
  Arms: Prednisolone 10; Prednisolone 60
Drug: Placebo
  Arms: Placebo

SUMMARY:
Although cortisone is widely used in the treatment of patients with early rheumatoid arthritis, the best dosage is not known. Therefore we will compare two standard prednisolon starting dosages and placebo in the treatment of patients with early active rheumatoid arthritis on the background of the established therapy with methotrexate. In total 450 patients will be included into the study. Two different treatment arms starting with 10 or 60 mg of prednisolone, and one placebo arm. Duration of intervention is 12 weeks. In parallel, all patients start medication with methotrexate, usual dosage 15 mg/week. Primary efficacy endpoint is progression of radiographic damage after one year compared to baseline. Safety monitoring is performed.

DETAILED DESCRIPTION:
BACKGROUND: Although glucocorticoids (GCs) are widely used in the treatment of patients with early rheumatoid arthritis (RA), the best dosage for GCs, related to both, efficacy and safety, is not known.

OBJECTIVE: To compare two standard p.o. GC starting dosages and the non-use of GCs in the treatment of patients with early active RA on the background of the established 'anchor' therapy with methotrexate (MTX).

METHODS: Randomised double-blind placebo-controlled trial with two treatment arms (starting with 10 or 60 mg of p.o. prednisolone (P), tapered down to 5 mg P per day within 8 weeks) and one placebo arm, each arm comprising 150 patients. Duration of intervention is 12 weeks. In parallel, all patients start medication with MTX, usual dosage 15 mg/week. Primary efficacy endpoint is progression of radiographic damage after one year compared to baseline. Secondary endpoints are: percentage of patients in remission, changes of functional capacity etc. Safety monitoring is performed.

The analysis is performed in three hierarchical steps. First step is an analysis of covariance to compare the group with an initial P dosage of 60 mg (V60) and the placebo group (Pl). In case of a statistical significant result (α = 0.05), a comparison of the group starting with 10 mg P (V10) and Pl will be done in a second step (α = 0.05). In case of superiority of V10 versus Pl, a third step will be a non-inferiority test for V10 versus V60 (α = 0.025).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis based on expert opinion according to the American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) 2009 criteria (Hawker 2009)
* disease duration < 3 years
* active disease: disease activity score (DAS) 28 erythrocyte sedimentation rate (ESR) (Prevoo et al 1995) > 4 plus ≥ 3 swollen joints

Exclusion Criteria:

* Prior treatment with disease-modifying antirheumatic drugs (DMARDs) (except for hydroxychloroquine or sulfasalazine or methotrexate during the last four weeks before screening)
* Clinically relevant comorbidity:
* concurrent liver disease (ALT > 2 times upper limit of normal),
* active hepatitis B or C viral infection,
* renal disease (creatinine clearance < 30 ml/minute),
* clinically relevant haematological disease due to the judgement of the rheumatologist,
* uncontrolled diabetes mellitus,
* uncontrolled arterial hypertension,
* relevant immunodeficiency incl. HIV-infection,
* clinically significant pulmonary fibrosis,
* history of malignant melanoma,
* complicated or refractory gastrointestinal ulcers,
* presence or history of severe infections,
* uncontrolled increased intraocular pressure,
* pregnancy or planned pregnancy,
* non-compliance,
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Progression of radiographic damage after one year as quantified by the van der Heijde modification of the Sharp score (SHS). Determined at baseline and after one year. | 52 weeks
  15 sites in each hand and wrist and six joints in each foot are examined for joint space narrowing on a scale of 0 to 437: 0 indicates no narrowing, 1 represents minimal narrowing, 2 indicates loss of 50% of the joint space, 3 indicates loss of 75% of the joint space, and 4 represents complete loss of the joint space. The erosions are counted individually, usually at 16 sites in each hand and wrist and six sites in each foot, with a maximum score of 5 given for a destroyed hand or foot joint. For joints in the feet, the van der Heijde version of the Sharp scoring system has a maximum score of 10 for a destroyed joint

SECONDARY OUTCOMES:
Percentage of patients in remission | 12 weeks, 24 weeks, 52 weeks
  as defined by the DAS 28 score
Changes of functional capacity | Baseline, 12 weeks, 52 weeks
  as defined by the so called "Hannover function questionnaire"
Patient's assessment of disease activity | Baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks, 52 weeks
  on a scale between 0 and 10

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Braun, MD, Principal Investigator — Rheumazentrum Ruhrgebiet, Herne/Germany
Locations (25):
- Germany (25):
  - Rheumatologische Schwerpunktpraxis Bielefeld, Bielefeld
  - Rheumatologische Schwerpunktpraxis Bocholt, Bocholt
  - Rheumatologische Schwerpunktpraxis Bochum, Bochum
  - Rheumaticon Internistische Schwerpunktpraxis Immunologie, Rheumatologie, Osteologie JosefCarrée Bochum, Bochum
  - Rheumapraxis Dortmund, Dortmund
  - MVZ Dr. Kretzmann und Kollegen, Dortmund
  - Rheumatologische Schwerpunktpraxis Dortmund, Dortmund
  - Rheumapraxis Duisburg, Duisburg
  - Rheumapraxis Gelsenkirchen, Gelsenkirchen
  - Internistische und rheumatologische Praxis Gladbeck, Gladbeck
  - Facharztzentrum Hagen, Hagen
  - Orthopädisch-rheumatologische Schwerpunktpraxis, Hattingen
  - Rheumapraxis Hattingen, Hattingen
  - Rheumazentrum Ruhrgebiet, Herne
  - Rheumapraxis Herne, Herne
  - Rheumatologische Schwerpunktpraxis Lingen, Lingen
  - Rheumapraxis am EVK, Lippstadt
  - Rheumatologische Schwerpunktpraxis Marl, Marl
  - Rheumatologische Schwerpunktpraxis Minden, Minden
  - Rheumatologische Schwerpunktpraxis Münster, Münster
  - Rheumapraxis Oberhausen, Oberhausen
  - Rheumapraxis Paderborn, Paderborn
  - Rheumazentrum Ratingen, Ratingen
  - Rheumatologische Schwerpunktpraxis Rheine, Rheine
  - Rheumapraxis Warendorf, Warendorf

REFERENCES:
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595
- [Background] Bakker MF, Jacobs JW, Welsing PM, Verstappen SM, Tekstra J, Ton E, Geurts MA, van der Werf JH, van Albada-Kuipers GA, Jahangier-de Veen ZN, van der Veen MJ, Verhoef CM, Lafeber FP, Bijlsma JW; Utrecht Rheumatoid Arthritis Cohort Study Group. Low-dose prednisone inclusion in a methotrexate-based, tight control strategy for early rheumatoid arthritis: a randomized trial. Ann Intern Med. 2012 Mar 6;156(5):329-39. doi: 10.7326/0003-4819-156-5-201203060-00004. PMID 22393128
- [Background] Bijlsma JW, van der Goes MC, Hoes JN, Jacobs JW, Buttgereit F, Kirwan J. Low-dose glucocorticoid therapy in rheumatoid arthritis: an obligatory therapy. Ann N Y Acad Sci. 2010 Apr;1193:123-6. doi: 10.1111/j.1749-6632.2009.05342.x. PMID 20398017
- [Background] Boers M, Verhoeven AC, Markusse HM, van de Laar MA, Westhovens R, van Denderen JC, van Zeben D, Dijkmans BA, Peeters AJ, Jacobs P, van den Brink HR, Schouten HJ, van der Heijde DM, Boonen A, van der Linden S. Randomised comparison of combined step-down prednisolone, methotrexate and sulphasalazine with sulphasalazine alone in early rheumatoid arthritis. Lancet. 1997 Aug 2;350(9074):309-18. doi: 10.1016/S0140-6736(97)01300-7. PMID 9251634
- [Background] Breedveld FC, Han C, Bala M, van der Heijde D, Baker D, Kavanaugh AF, Maini RN, Lipsky PE. Association between baseline radiographic damage and improvement in physical function after treatment of patients with rheumatoid arthritis. Ann Rheum Dis. 2005 Jan;64(1):52-5. doi: 10.1136/ard.2003.017160. Epub 2004 Jul 29. PMID 15286005
- [Background] Capell HA, Madhok R, Hunter JA, Porter D, Morrison E, Larkin J, Thomson EA, Hampson R, Poon FW. Lack of radiological and clinical benefit over two years of low dose prednisolone for rheumatoid arthritis: results of a randomised controlled trial. Ann Rheum Dis. 2004 Jul;63(7):797-803. doi: 10.1136/ard.2003.014050. PMID 15194574
- [Background] Choy EH, Smith CM, Farewell V, Walker D, Hassell A, Chau L, Scott DL; CARDERA (Combination Anti-Rheumatic Drugs in Early Rheumatoid Arhritis) Trial Group. Factorial randomised controlled trial of glucocorticoids and combination disease modifying drugs in early rheumatoid arthritis. Ann Rheum Dis. 2008 May;67(5):656-63. doi: 10.1136/ard.2007.076299. Epub 2007 Sep 3. PMID 17768173
- [Background] Goekoop-Ruiterman YP, de Vries-Bouwstra JK, Allaart CF, van Zeben D, Kerstens PJ, Hazes JM, Zwinderman AH, Ronday HK, Han KH, Westedt ML, Gerards AH, van Groenendael JH, Lems WF, van Krugten MV, Breedveld FC, Dijkmans BA. Clinical and radiographic outcomes of four different treatment strategies in patients with early rheumatoid arthritis (the BeSt study): a randomized, controlled trial. Arthritis Rheum. 2005 Nov;52(11):3381-90. doi: 10.1002/art.21405. PMID 16258899
- [Background] Grigor C, Capell H, Stirling A, McMahon AD, Lock P, Vallance R, Kincaid W, Porter D. Effect of a treatment strategy of tight control for rheumatoid arthritis (the TICORA study): a single-blind randomised controlled trial. Lancet. 2004 Jul 17-23;364(9430):263-9. doi: 10.1016/S0140-6736(04)16676-2. PMID 15262104
- [Background] Gorter SL, Bijlsma JW, Cutolo M, Gomez-Reino J, Kouloumas M, Smolen JS, Landewe R. Current evidence for the management of rheumatoid arthritis with glucocorticoids: a systematic literature review informing the EULAR recommendations for the management of rheumatoid arthritis. Ann Rheum Dis. 2010 Jun;69(6):1010-4. doi: 10.1136/ard.2009.127332. Epub 2010 May 6. PMID 20448288
- [Background] Hoes JN, Jacobs JW, Verstappen SM, Bijlsma JW, Van der Heijden GJ. Adverse events of low- to medium-dose oral glucocorticoids in inflammatory diseases: a meta-analysis. Ann Rheum Dis. 2009 Dec;68(12):1833-8. doi: 10.1136/ard.2008.100008. Epub 2008 Dec 9. PMID 19066177
- [Background] Hoes JN, Jacobs JW, Buttgereit F, Bijlsma JW. Current view of glucocorticoid co-therapy with DMARDs in rheumatoid arthritis. Nat Rev Rheumatol. 2010 Dec;6(12):693-702. doi: 10.1038/nrrheum.2010.179. PMID 21119718
- [Background] Kirwan JR. The effect of glucocorticoids on joint destruction in rheumatoid arthritis. The Arthritis and Rheumatism Council Low-Dose Glucocorticoid Study Group. N Engl J Med. 1995 Jul 20;333(3):142-6. doi: 10.1056/NEJM199507203330302. PMID 7791815
- [Background] Mottonen T, Hannonen P, Leirisalo-Repo M, Nissila M, Kautiainen H, Korpela M, Laasonen L, Julkunen H, Luukkainen R, Vuori K, Paimela L, Blafield H, Hakala M, Ilva K, Yli-Kerttula U, Puolakka K, Jarvinen P, Hakola M, Piirainen H, Ahonen J, Palvimaki I, Forsberg S, Koota K, Friman C. Comparison of combination therapy with single-drug therapy in early rheumatoid arthritis: a randomised trial. FIN-RACo trial group. Lancet. 1999 May 8;353(9164):1568-73. doi: 10.1016/s0140-6736(98)08513-4. PMID 10334255
- [Background] Mouterde G, Dernis E, Ruyssen-Witrand A, Claudepierre P, Schaeverbeke T, Cantagrel A, Gaudin P, Maillefert JF, Pham T, Saraux A, Tebib J, Wendling D, Fautrel B, Le Loet X. Indications of glucocorticoids in early arthritis and rheumatoid arthritis: recommendations for clinical practice based on data from the literature and expert opinion. Joint Bone Spine. 2010 Dec;77(6):597-603. doi: 10.1016/j.jbspin.2009.12.011. Epub 2010 Jul 1. PMID 20594896
- [Background] Smolen JS, Aletaha D, Bijlsma JW, Breedveld FC, Boumpas D, Burmester G, Combe B, Cutolo M, de Wit M, Dougados M, Emery P, Gibofsky A, Gomez-Reino JJ, Haraoui B, Kalden J, Keystone EC, Kvien TK, McInnes I, Martin-Mola E, Montecucco C, Schoels M, van der Heijde D; T2T Expert Committee. Treating rheumatoid arthritis to target: recommendations of an international task force. Ann Rheum Dis. 2010 Apr;69(4):631-7. doi: 10.1136/ard.2009.123919. Epub 2010 Mar 9. PMID 20215140
- [Background] Smolen JS, Landewe R, Breedveld FC, Dougados M, Emery P, Gaujoux-Viala C, Gorter S, Knevel R, Nam J, Schoels M, Aletaha D, Buch M, Gossec L, Huizinga T, Bijlsma JW, Burmester G, Combe B, Cutolo M, Gabay C, Gomez-Reino J, Kouloumas M, Kvien TK, Martin-Mola E, McInnes I, Pavelka K, van Riel P, Scholte M, Scott DL, Sokka T, Valesini G, van Vollenhoven R, Winthrop KL, Wong J, Zink A, van der Heijde D. EULAR recommendations for the management of rheumatoid arthritis with synthetic and biological disease-modifying antirheumatic drugs. Ann Rheum Dis. 2010 Jun;69(6):964-75. doi: 10.1136/ard.2009.126532. Epub 2010 May 5. PMID 20444750
- [Background] Sokka T, Abelson B, Pincus T. Mortality in rheumatoid arthritis: 2008 update. Clin Exp Rheumatol. 2008 Sep-Oct;26(5 Suppl 51):S35-61. PMID 19026144
- [Background] Svensson B, Boonen A, Albertsson K, van der Heijde D, Keller C, Hafstrom I. Low-dose prednisolone in addition to the initial disease-modifying antirheumatic drug in patients with early active rheumatoid arthritis reduces joint destruction and increases the remission rate: a two-year randomized trial. Arthritis Rheum. 2005 Nov;52(11):3360-70. doi: 10.1002/art.21298. PMID 16255010
- [Background] van der Goes MC, Jacobs JW, Boers M, Andrews T, Blom-Bakkers MA, Buttgereit F, Caeyers N, Cutolo M, Da Silva JA, Guillevin L, Kirwan JR, Rovensky J, Severijns G, Webber S, Westhovens R, Bijlsma JW. Monitoring adverse events of low-dose glucocorticoid therapy: EULAR recommendations for clinical trials and daily practice. Ann Rheum Dis. 2010 Nov;69(11):1913-9. doi: 10.1136/ard.2009.124958. Epub 2010 Aug 6. PMID 20693273
- [Background] van Everdingen AA, Jacobs JW, Siewertsz Van Reesema DR, Bijlsma JW. Low-dose prednisone therapy for patients with early active rheumatoid arthritis: clinical efficacy, disease-modifying properties, and side effects: a randomized, double-blind, placebo-controlled clinical trial. Ann Intern Med. 2002 Jan 1;136(1):1-12. doi: 10.7326/0003-4819-136-1-200201010-00006. PMID 11777359
- [Background] van Vollenhoven RF, Cifaldi MA, Ray S, Chen N, Weisman MH. Improvement in work place and household productivity for patients with early rheumatoid arthritis treated with adalimumab plus methotrexate: work outcomes and their correlations with clinical and radiographic measures from a randomized controlled trial companion study. Arthritis Care Res (Hoboken). 2010 Feb;62(2):226-34. doi: 10.1002/acr.20072. PMID 20191522
- [Background] Wassenberg S, Rau R, Steinfeld P, Zeidler H. Very low-dose prednisolone in early rheumatoid arthritis retards radiographic progression over two years: a multicenter, double-blind, placebo-controlled trial. Arthritis Rheum. 2005 Nov;52(11):3371-80. doi: 10.1002/art.21421. PMID 16255011
- [Background] Wolfe F, Michaud K. The risk of myocardial infarction and pharmacologic and nonpharmacologic myocardial infarction predictors in rheumatoid arthritis: a cohort and nested case-control analysis. Arthritis Rheum. 2008 Sep;58(9):2612-21. doi: 10.1002/art.23811. PMID 18759273
- [Background] Dachverband Osteologie e.V., DVO-Leitlinie 2009 zur Prophylaxe, Diagnostik und Therapie der Osteoporose bei Erwachsenen, Osteologie 4/2009: 304 -324.
- [Derived] Trampisch US, Krause D, Trampisch HJ, Klaassen-Mielke R, Baraliakos X, Braun J. Comparison of the efficacy and safety of two starting dosages of prednisolone in early active rheumatoid arthritis (CORRA): study protocol for a randomized controlled trial. Trials. 2014 Sep 2;15:344. doi: 10.1186/1745-6215-15-344. PMID 25181946